CLINICAL TRIAL: NCT05263622
Title: Guided Biofilm Therapy for Periodontal Patients Using Two Different Devices: a Split-mouth Randomized Clinical Trial
Brief Title: Guided Biofilm Therapy for Periodontal Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-GBT
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Periodontal Diseases
Keywords: Guided Biofilm Therapy
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Split-mouth design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Half of patients will be included in this group according to the split-mouth design.
  Interventions: Other: Split-mouth administration for group A
- Group B (Experimental): Half of patients will be included in this group according to the split-mouth design.
  Interventions: Other: Split-mouth administration for group B

INTERVENTIONS:
Other: Split-mouth administration for group B — * Plaque disclosing agent application and instructions to patients for a correct oral hygiene;
  * Airflow deplaquing with EMS handpiece (quadrants Q1 and Q3) and with Mectron handpiece (quadrants Q2 and Q4)
  * Calculus removal with EMS ultrasound handpiece (Q1 and Q3) and with Mectron handpiece (Q2 and Q4)
  Arms: Group B
Other: Split-mouth administration for group A — * Plaque disclosing agent application and instructions to patients for a correct oral hygiene;
  * Airflow deplaquing with EMS handpiece (quadrants Q2 and Q4) and with Mectron handpiece (quadrants Q1 and Q3)
  * Calculus removal with EMS ultrasound handpiece (Q2 and Q4) and with Mectron handpiece (Q1 and Q3)
  Arms: Group A

SUMMARY:
Periodontal patients will be treated with Guided Biofilm Therapy. At the baseline (T0), the following clinical indices will be collected: BoP, BS, CAL, PPD. A plaque disclosing agents will be used to instruct the patients to proper oral hygiene procedures. At this stage, using a split-mouth design, quadrants will be randomized to:

* Airflow and Scaling and calculus removal with EMS Prophylaxis Master handpiece
* Airflow and calculus removal with Mectron Combi handpiece

Patients will be visited after 1 month (T1) and 2 months (T2), in which the periodontal indexes will be collected again.

After all the procedures, VAS for pain will be assessed, with Schiff Air Index, comfort (patients), comfort (operator), timing for the procedures (minutes), satisfaction questionnaire (for patients and for the operator), consumption of the powders for the two handpiece.

DETAILED DESCRIPTION:
Periodontal patients that respond to the inclusion criteria and agree to participate in the study will be treated with Guided Biofilm Therapy.

At the baseline (T0), the following clinical indices will be collected: BoP, BS, CAL, PPD. A plaque disclosing agents will be used to instruct the patients to proper oral hygiene procedures. At this stage, using a split-mouth design, quadrants will be randomized to:

* Airflow and calculus removal with EMS Prophylaxis Master handpiece
* Airflow and calculus removal with Mectron Combi handpiece

Patients will be visited after 1 month (T1) and 2 months (T2), in which the periodontal indexes will be collected again.

Together with periodontal assessment, VAS for pain will be assessed, with Schiff Air Index, comfort (patients), comfort (operator), timing for the procedures (minutes), satisfaction questionnaire (for patients and for the operator), consumption of the powders for the two handpieces.

ELIGIBILITY:
Inclusion Criteria:

* professional dental hygiene performed at least 6 months before enrollment
* periodontal disease: grading A or B and staging I-III

Exclusion Criteria:

* neurologic, psychiatric and mental diseases
* patients taking antibiotics during the study
* pregnant and breastfeeding women
* patients undergoing anticancer treatment
* patients undergoing anticancer therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Change in Schiff Air Index - Dental sensitivity test | Baseline, after 30 and 60 days
  Scoring criteria:
  0. the subject did not respond to air blasting;
  1. the subject responded to air blasting;
  2. the subject responded to air blasting and requested discontinuation;
  3. the subject responded to air blasting, requested discontinuation and considered the stimulus to be painful.
Change in BOP - Bleeding on Probing (percentage) | Baseline, after 30 and 60 days
  Site-specific assessment of the presence or absence of gum bleeding after the insertion of the periodontal probe for the detection of PPD, detected on 4 sites (mesial, distal, vestibular, palatal/lingual).
Change in Bleeding Score (BS - Mombelli et al.) | Baseline, after 30 and 60 days
  Scoring criteria:
  0: no bleeding
  1. isolated visible spots
  2. blood forms a confluent red line on the mucosal margin
  3. profuse and copious bleeding
Change in Probing Pocket Depth (PPD) | Baseline, after 30 and 60 days
  Evaluation (in mm) of the depth of the gingival sulcus, through a millimeter periodontal probe; it is detected from the gingival margin to the bottom of the gingival sulcus or periodontal pocket, evaluated at 6 sites.
Change in CAL - Clinical Attachment Loss | Baseline, after 30 and 60 days
  Measurement (in mm) of the position of the gingival margin in relation to the cemento-enamel junction (CEJ).
Total time of usage | Baseline
  Total time of usage of the two handpieces.
Comfort for the operator | Baseline
  Evaluation of the comfort of the operator from 0 to 10 during professional procedures.
Satisfactory questionnaire for patients | Baseline
  Choice of a score from 0 to 10 for all the following questions:
  * Is the time for the procedures appropriate?
  * Is the quantity of droplets adequate?
  * Dental sensitivity
  * Pain with the first instrument
  * Pain with the second instrument
  * General pain
Satisfactory questionnaire for operator | Baseline
  Comfort (from 0 to 10) Timing (from 0 to 10)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, MS, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

REFERENCES:
- [Derived] Chiesa A, Pascadopoli M, Butera A, Monticone M, Mirando M, Vezzoni F, Kertalli A, Scribante A, Nardi GM. Differences Between Two Devices With Function of Periopolishing and Piezoelectric Scaler: A Randomized Clinical Trial. Int J Dent. 2025 Mar 4;2025:7131637. doi: 10.1155/ijod/7131637. eCollection 2025. PMID 40223867